CLINICAL TRIAL: NCT04018547
Title: Investigating the Use of a Wrist-sensor Pulse Oximeter to Screen for Obstructive Sleep Apnoea.
Brief Title: Investigating a Wrist-sensor Oximeter to Screen for Sleep Apnoea.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oxitone Medical Ltd. (Industry)
Collaborators: The London Sleep Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 265604
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Screening, patient convenience
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Patient wears a wrist sensor oximeter device for one to two nights. — Patients will be asked to complete a study questionnaires of STOPBANG, SCI-8 (Sleep Condition Indicator-8 questionnaire for insomnia), Epworth questionnaires and medical history. The clinician will record blood pressure, pulse rate and regularity, body mass index and neck circumference. Subjects will be required to wear the wrist sensor pulse oximeter for 1-2 nights. The Oxitone 1000M device measures pulse rate, blood oxygen saturation and movement. The oxygen desaturation events from the wrist sensor device will be statistically compared with the diagnosis assessed using the conventional PPG oximetry, Peripheral Arterial Tonometry and clinical assessment. (clinicians will be masked when analysing the data from the wrist sensor pulse device).

SUMMARY:
The primary study objective is to investigate sensitivity and specificity of a wrist sensor pulse oximeter (the Oxitone Medical Oxitone 1000M device) to screen for obstructive sleep apnoea. This study will involve thirty participants attending a sleep centre suspected of suffering from obstructive sleep apnoea (case finding screening). The secondary objective is to assess patient convenience with the screening procedure.

DETAILED DESCRIPTION:
This is an observational study to assess the sensitivity and specificity of a wrist sensor pulse oximeter (Oxitone Medical Oxitone 1000M) to identify obstructive sleep apnoea cases in patients referred to the London Sleep Centre (case finding screening, or case only study). The wrist sensor pulse oximeter streams data (pulse rate, heart rate variability (HRV), blood oxygen saturation levels (SPO2), actigraphy data and skin temperature data) to a software application using bluetooth connectivity to be stored in a securely encrypted database cloud for analysis. The investigators at the sleep centre will be masked when analysing the data from the wrist sensor pulse oximeter when deciding on diagnosis of obstructive sleep apnoea. Data from the wrist sensor oximeter device will be statistically compared with the data from a conventional PPG fingertip oximeter and Peripheral Arterial Tonometry device currently in use. The study outcome will be whether the wrist sensor pulse oximeter device could be used in patients to screen reliably for obstructive sleep apnoea. The study also will include patient feedback on convenience of the screening procedure. The study will not affect routine patient medical management and care for patients assessed at the sleep centre.

ELIGIBILITY:
Inclusion Criteria:

* Thirty consecutive patients referred to the sleep Centre for screening for sleep apnoea that consented to involvement in the study.

Exclusion Criteria:

* Patients who are unable to give written informed consent.
* anaemia or dysfunctional hemoglobin
* upper limb complaints affecting the ability to wear the watch like wrist sensor device such as tenderness, deformity or swelling, skin complaints such as ulceration, swelling or skin breaks
* impairment in circulation in the left upper limb (active Raynauds or other vascular impairment)
* neurological conditions such as tremor or convulsions
* Medical conditions likely to affect the blood oxygen such as chronic obstructive pulmonary disease (COPD) and chronic asthma
* Neurological conditions likely to affect breathing such as stroke
* Conditions likely to affect autonomic nervous system such as diabetes mellitus

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty consecutive patients referred to the sleep Centre for screening for sleep apnoea that consented to involvement in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-17 (Estimated); Primary Completion 2019-12-17 (Estimated); Study Completion 2019-12-17 (Estimated)

PRIMARY OUTCOMES:
obstructive sleep apnoea screening | Three months
  Sensitivity and specificity of the wrist sensor oximeter to screen for obstructive sleep apnoea by (A) comparing the SPO2 3% and 4 % dip rates of the conventional fingertip photoplethysmography(PPG) oximeter to the 3% and 4% dip rates of the wrist sensor pulse oximeter and (B) comparing the final diagnosis of obstructive sleep apnoea (OSA) by a sleep specialist (based on PPG fingertip oximetry and peripheral arterial tonometry), with SPO2 and heart rate variability data from the wrist sensor pulse oximeter. The sleep specialist will be masked from the data of the wrist sensor pulse oximeter. An ROC (receiver operating characteristic) curve will be used for (B).

SECONDARY OUTCOMES:
Patient comfort and compliance | Three months
  To assess patient comfort wearing the wrist sensor pulse oximetry device by administering a questionnaire with responses on a Likert scale to question "the wrist sensor pulse oximeter was comfortable to sleep with"

CONTACTS AND LOCATIONS:
Locations (1):
- London Sleep Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared with other researchers.
  Personal identifiable data will not be shared with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: Three months
Access Criteria: Contact Oxitone for access
URL: http://www.oxitone.com

REFERENCES:
- Available data/document: Individual Participant Data Set — http://www.oxitone.com — De-identified data for primary and secondary outcome measures